CLINICAL TRIAL: NCT00231023
Title: Pilot Study of Peribulbar Triamcinolone Acetonide for Diabetic Macular Edema
Brief Title: Triamcinolone Acetonide Injections to Treat Diabetic Macular Edema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050251; 05-EI-0251
Record Dates: First submitted 2005-10-02; First posted 2005-10-03 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-05

CONDITIONS: Diabetic Retinopathy
Keywords: Anterior Subtenon; Posterior Peribulbar; Laser Photocoagulation; Diabetes; Diabetic Retinopathy; Diabetic Macular Edema; DME
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus

INTERVENTIONS:
Drug: Peribulbar Triamcinolone Acetonide

SUMMARY:
This study will evaluate which of the three following treatment options is better for diabetic macular edema: laser alone, steroid injection alone, or steroid injection followed by laser. Macular edema is a swelling in the small central part of the retina - the part of the retina that is used for sharp, straight-ahead vision. Laser treatment is the only treatment that has been proven to be beneficial for diabetic macular edema. It reduces the swelling and lessens the chance of further vision loss, but it does not improve vision. Triamcinolone is a steroid drug that decreases inflammation and scarring. Injections of the drug have decreased macular edema in some patients and improved vision. Swelling may return, requiring repeat injections, and it is not known if the vision improvement is permanent. This 3-year study will examine and compare the benefits and side effects of both treatments, alone and in combination.

Patients 18 years of age and older with diabetic macular edema may be eligible for this study. Participants undergo the following tests and procedures.

At the beginning of the study:

* Blood tests to measure HbA1C (measure of diabetes control).
* Measurement of blood pressure.
* Eye examination to assess visual acuity (eye chart test) and eye pressure, and to examine pupils, lens, retina and eye movements. The pupils are dilated with drops for this examination.
* Optical coherence tomography (OCT) to measure retinal thickness. This test shines a light into the eye and produces cross-sectional pictures of the retina. These measurements are repeated during the study to determine if retinal thickening is getting better or worse, or staying the same.

Photographs of the retina and lens. A special camera with bright flashes is used to take these photographs.

Treatments

Some patients will have one eye treated and some patients will have both eyes treated. The treatment for a given individual is determined by chance:

* Triamcinolone acetonide injection alone. The steroid is injected in the tissue around the eye. Two injection procedures are used in the study, differing in their location and dose. Numbing drops are placed over the area to be injected and the steroid is injected.
* Laser treatment alone. The surface of the eye is numbed with drops and a contact lens is placed on the eye during the laser beam application. Before the treatment, patients may have fluorescein angiography, in which pictures of the retina are taken using a yellow dye. The dye is injected into a vein and travels to the blood vessels in the eye. The camera flashes a blue light in the eye and takes pictures that show the amount of dye leakage into the retina. Treatments may be repeated at several visits.
* Triamcinolone acetonide plus laser treatment. Patients who receive both the steroid injection and laser have the steroid injection first and the laser treatment 1 month later.

Follow-up

Patients return to the clinic for follow-up visits at 1, 2, 4, 8, 12, 24 and 36 months, or more often if needed, after the initial treatment for an eye exam, measurement of visual acuity, and OTC. Photographs of the retina are taken at the 4- and 8-month visits and at the 1-, 2- and 3-year visits. Fluorescein angiography may be done at 4 months. Blood pressure is measured at the 1-, 2- and 3-year visits, and an HbA1c blood test is done at 4 and 8 months and at the yearly visits. Participants may be asked to complete a questionnaire once a year about their vision and medical condition. Treatment options are discussed at the 4- and 8-month visits.

DETAILED DESCRIPTION:
Diabetic retinopathy is a major cause of visual impairment in the United States. Diabetic macular edema (DME) is a manifestation of diabetic retinopathy that produces loss of central vision. Data from the Wisconsin Epidemiologic Study of Diabetic Retinopathy (WESDR) estimate that after 15 years of known diabetes, the prevalence of diabetic macular edema is approximately 20% in patients with type 1 diabetes mellitus (DM), 25% in patients with type 2 DM who are taking insulin, and 14% in patients with type 2 DM who do not take insulin.

In a review of three early studies concerning the natural history of diabetic macular edema, Ferris and Patz found that 53% of 135 eyes with diabetic macular edema, presumably all involving the center of the macula, lost two or more lines of visual acuity over a two year period. In the Early Treatment Diabetic Retinopathy Study (ETDRS), 33% of 221 untreated eyes available for follow-up at the 3-year visit, all with edema involving the center of the macula at baseline, had experienced a 15 or more letter decrease in visual acuity score (equivalent to a doubling of the visual angle, e.g., 20/25 to 20/50, and termed "moderate visual loss").

In the ETDRS, focal/grid photocoagulation of eyes with clinically significant macular edema (CSME) reduced the risk of moderate visual loss by approximately 50% (from 24% to 12%, three years after initiation of treatment). Therefore, 12% of treated eyes developed moderate visual loss in spite of treatment. Furthermore, approximately 40% of treated eyes that had retinal thickening involving the center of the macula at baseline still had thickening involving the center at 12 months, as did 25% of treated eyes at 36 months.

Although several treatment modalities are currently under investigation, the only demonstrated means to reduce the risk of vision loss from diabetic macular edema are laser photocoagulation, as demonstrated by the ETDRS, and intensive glycemic control, as demonstrated by the Diabetes Control and Complications Trial (DCCT) and the United Kingdom Prospective Diabetes Study (UKPDS). In the DCCT, intensive glucose control reduced the risk of onset of diabetic macular edema by 23% compared with conventional treatment. Long-term follow-up of patients in the DCCT show a sustained effect of intensive glucose control, with a 58% risk reduction in the development of diabetic macular edema for the DCCT patients followed in the Epidemiology of Diabetes Interventions and Complications Study.

The frequency of an unsatisfactory outcome following laser photocoagulation in some eyes with diabetic macular edema has prompted interest in other treatment modalities. One such treatment is pars plana vitrectomy. These studies suggest that vitreomacular traction, or the vitreous itself, may play a role in increased retinal vascular permeability. Removal of the vitreous or relief of mechanical traction with vitrectomy and membrane stripping may be followed by substantial resolution of macular edema and corresponding improvement in visual acuity. However, this treatment may be applicable only to a specific subset of eyes with diabetic macular edema. It also requires a complex surgical intervention with its inherent risks, recovery time, and expense. Other treatment modalities such as pharmacologic therapy with oral protein kinase C inhibitors and antibodies targeted at vascular endothelial growth factor (VEGF) are under investigation.

The use of intravitreal corticosteroids is another treatment modality that has generated recent interest. However, use of intravitreal corticosteroids generally has been reserved for cases of DME in which there is at least moderate loss of visual acuity (e.g., worse than 20/40). This treatment generally has not been widely used for mild cases of DME due to concerns about its potential risks, particularly glaucoma and cataract, relative to the potential benefit.

Injection of corticosteroids around the eye (anterior subtenon's, posterior subtenon's, retrobulbar) has been used as an alternative to intravitreal injection. Although data are limited, it is presumed that the adverse effects on the eye are lower with an injection around the eye compared with in the eye. There are also little data on the efficacy of this treatment. This study is being conducted to collect pilot data on the safety and efficacy of peribulbar corticosteroids to determine whether there is sufficient evidence of efficacy to merit conducting a phase 3 randomized trial.

ELIGIBILITY:
SUBJECT-LEVEL CRITERIA

INCLUSION CRITERIA

To be eligible, the following inclusion criteria (1-4) must be met:

-Age greater than or equal to 18 years

1. Patients less than18 years old are not being included because DME is so rare in this age group that the diagnosis of DME may be questionable.
2. Diagnosis of diabetes mellitus (type 1 or type 2)

   - Any one of the following will be considered to be sufficient evidence that diabetes is present:

   Current regular use of insulin for the treatment of diabetes

   Current regular use of oral anti-hyperglycemia agents for the treatment of diabetes

   Documented diabetes by ADA and/or WHO criteria
3. At least one eye meets the study eye criteria
4. Able and willing to provide informed consent.

EXCLUSION

A patient is not eligible if any of the following exclusion criteria (5-13) are present:

5. History of chronic renal failure requiring dialysis or kidney transplant.

6. A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure and glycemic control).

* Patients in poor glycemic control who, within the last 4 months, initiated intensive insulin treatment (a pump or multiple daily injections) or plan to do so in the next 4 months should not be enrolled.

  7. Participation in an investigational trial within 30 days of study entry that involved treatment with any drug that has not received regulatory approval at the time of study entry.

  8. Known allergy to any corticosteroid or any component of the delivery vehicle.

  9. History of systemic (e.g., oral, IV, IM, epidural, bursal) corticosteroids within 4 months prior to randomization or topical, rectal, or inhaled corticosteroids in current use more than 2 times per week.

  10. History of steroid-induced intraocular pressure elevation that required IOP-lowering treatment in either eye.

  11. Warfarin (coumadin) currently being used.

  12. Blood pressure greater than 180/110 (systolic above 180 OR diastolic above 110).
* If blood pressure is brought below 180/110 by anti-hypertensive treatment, patient can become eligible.

  13. Patient is expecting to move out of the area of the clinical center to an area not covered by another clinical center during the next 8 months.

STUDY EYE CRITERIA

The patient must have at least one eye meeting all of the inclusion criteria (a-e) and none of the exclusion criteria (f-t) listed below.

A patient may have two study eyes only if both are eligible at the time of randomization

The eligibility criteria for a study eye are as follows:

INCLUSION CRITERIA

1. Best corrected E-ETDRS visual acuity score of greater than or equal to 69 letters (i.e., 20/40 or better).
2. Definite retinal thickening due to diabetic macular edema based on clinical exam.
3. Retinal thickness in the OCT central subfield measuring 250 microns or more
4. Maximal laser has not already been given and investigator believes that either peribulbar steroids or laser may benefit the eye (note: subjects may be enrolled without having received prior macular laser).
5. Media clarity, pupillary dilation, and patient cooperation sufficient for adequate fundus photographs and OCT.

   EXCLUSION CRITERIA
6. Macular edema is considered to be due to a cause other than diabetic macular edema.

   - An eye should not be considered eligible: (1) if the macular edema is considered to be related to intraocular surgery such as cataract surgery or (2) clinical exam and/or OCT suggests that vitreoretinal interface abnormality (e.g., a taut posterior hyaloid or epiretinal membrane) is judged to be a cause of the macular edema.
7. An ocular condition is present such that, in the opinion of the investigator, visual acuity would not improve from resolution of macular edema (e.g., foveal atrophy, pigmentary changes, dense subfoveal hard exudates, nonretinal condition).
8. An ocular condition is present (other than diabetes) that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the course of the study (e.g., vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, Irvine-Gass Syndrome, etc.).
9. History of prior treatment with intravitreal, peribulbar, or retrobulbar corticosteroids for DME.
10. History of focal/grid macular photocoagulation within 15 weeks (3.5 months) prior to randomization.

    - Note: Patients are not required to have had prior macular photocoagulation to be enrolled.
11. History of panretinal scatter photocoagulation (PRP) within 4 months prior to randomization.
12. Anticipated need for PRP in the 4 months following randomization.
13. History of prior vitrectomy.
14. History of major ocular surgery (including cataract extraction, scleral buckle, any intraocular surgery, etc.) within prior 6 months or anticipated within the next 6 months following randomization.
15. History of YAG capsulotomy performed within 2 months prior to randomization.
16. Intraocular pressure greater than or equal to 25 mmHg.
17. History of open-angle glaucoma (either primary open-angle glaucoma or other cause of open-angle glaucoma; note: angle-closure glaucoma is not an exclusion).

    * A history of ocular hypertension is not an exclusion as long as (1) intraocular pressure is less than 25 mm Hg, (2) the patient is using no more than one topical glaucoma medication, (3) the most recent visual field, performed within the last 12 months, is normal (if abnormalities are present on the visual field they must be attributable to the patient's diabetic retinopathy), and (4) the optic disc does not appear glaucomatous.
    * Note: if the intraocular pressure is 22 to less than 25 mm Hg, then the above criteria for ocular hypertension eligibility must be met.
18. History of prior herpetic ocular infection.
19. Exam evidence of ocular toxoplasmosis.
20. Exam evidence of pseudoexfoliation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10
Dates: Start 2005-09; Study Completion 2006-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Eye Institute (NEI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Klein R, Klein BE, Moss SE, Davis MD, DeMets DL. The Wisconsin epidemiologic study of diabetic retinopathy. IV. Diabetic macular edema. Ophthalmology. 1984 Dec;91(12):1464-74. doi: 10.1016/s0161-6420(84)34102-1. PMID 6521986
- [Background] Moss SE, Klein R, Klein BE. Ten-year incidence of visual loss in a diabetic population. Ophthalmology. 1994 Jun;101(6):1061-70. doi: 10.1016/s0161-6420(94)31217-6. PMID 8008348
- [Background] Moss SE, Klein R, Klein BE. The 14-year incidence of visual loss in a diabetic population. Ophthalmology. 1998 Jun;105(6):998-1003. doi: 10.1016/S0161-6420(98)96025-0. PMID 9627648